CLINICAL TRIAL: NCT00988533
Title: An Open-label Study to Assess the Bioavailability, Safety, Local Tolerance, and Efficacy of 0.5% Ivermectin Cream in Subjects 6 Months to 3 Years of Age With Pediculus Humanus Capitis (Head Lice) Infestation
Brief Title: A Pharmacokinetics (PK) Study in Lice Infested Children 6 Months to 3 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Topaz Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOP008
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2012-04-25 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-03

CONDITIONS: Head Lice
Keywords: Head Lice; Pediculus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.5% Ivermectin Cream (Experimental)
  Interventions: Drug: 0.5% Ivermectin Cream

INTERVENTIONS:
Drug: 0.5% Ivermectin Cream — Topical 0.5% ivermectin cream applied to scalp and hair on day 1

SUMMARY:
The purpose of this study is to determine the bioavailability of 0.5% ivermectin cream in a pediatric population aged 6 months to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 6 months to 3 years of age, inclusive, when informed consent is signed.
* Subject must be infested with head lice as demonstrated by the presence of at least 1 live louse prior to treatment.
* Subject is in general good health.
* Subject's parent/guardian (caregiver) must be willing and able to bring subject to all study visits as scheduled.
* Subject's caregiver must have provided written informed consent (assent is not required due to the young age of the subjects).
* Subject's caregiver must agree to comply with the following study restrictions:

  * will not use any other form of lice treatment (eg, commercial, community/anecdotal, or mechanical/manual) on the subject for the duration of the study, unless directed to do so by study personnel.
  * will not shampoo, wash, or rinse the subject's hair or scalp until the Day 2 treatment evaluation has been completed.
  * will not cut or chemically treat subject's hair in the period between screening and follow-up on Day 15.
  * will use only study-provided shampoo on the subject for the duration of the study.
  * will follow all study instructions.

Exclusion Criteria:

* Subjects who have received any OTC or prescription treatment for head lice in the last 2 weeks.
* Subjects or subjects' caregivers who are unable to comply with the study obligations and all study visits.
* Subjects whose caregivers do not understand the requirements for participation and/or may be likely to exhibit poor compliance, in the opinion of the Investigator.
* Subjects with eczema, atopic dermatitis, or other chronic conditions of the scalp and skin.
* Subjects with visible skin/scalp condition(s) that are not attributable to head lice infestation, such as an erythema score that is > 2, blisters, or any other condition that, in the opinion of the investigative personnel or Sponsor, would interfere with the PK, safety and/or efficacy evaluations.
* Subjects with a history of allergy to ivermectin or any ingredients commonly included in hair products such as shampoos, hair conditioners, or styling aids.
* Subjects with other diagnoses that, in the opinion of the Investigator, would interfere with the PK, safety, and/or efficacy assessments or would preclude study participation.
* Subjects who have been treated with a systemic antibiotic within 2 weeks before screening.
* Subject currently taking warfarin sodium (Coumadin®) or has taken within 2 weeks before screening.
* Subjects who have been enrolled in any clinical study within the past 30 days; subjects may not participate in another study while participating in this study.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Topaz
Locations (5):
- United States (5):
  - Children's Investigational Research Program, Bentonville, Arkansas
  - Universal BioPharma Research, Inc, Dinuba, California
  - Impact Clinical Trials, Los Angeles, California
  - Lice Source Solutions Inc, Plantation, Florida
  - Spence Medical Research L.L.C, Picayune, Mississippi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and treated from 22 September 2009 to 18 November 2009 at 3 US clinical centers.
Pre-assignment Details: A total of 30 participants who met the inclusion and exclusion criteria were enrolled and treated.
Groups:
- 0.5% Ivermectin: Participants received a single application of 0.5% ivermectin on Day 1.
Period: Overall Study
Arm/Group | 0.5% Ivermectin
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: Months] | 25.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 7
Region of Enrollment [Number; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Concentration of Ivermectin in Samples Collected Before Application and at Specified Post-Application Time Points
Description: Plasma concentrations of ivermectin were measured by validated and appropriate bioanalytical instruments and methods with a sensitivity of 0.05 ng/mL before application and on Day 1 (0.5, 1, and 6 hours), Day 2 (24 hours post-application), Day 8 (7 days post-application), and Day 15 (14 days post-application).
Time Frame: Before; 0.5, 1, 6, 24 hours and Up to 14 days post-application
Population: Plasma concentrations of Ivermectin were assessed in the pharmacokinetic (PK) population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 20
ng/mL
  0 Hour (N = 20) | 0.00000 (0.00000) [lower limit 0.00000]
  0.5 Hour (N = 19) | 0.02528 (0.11018) [lower limit 0.11018]
  1 Hour (N = 19) | 0.08192 (0.22695) [lower limit 0.22695]
  6 Hours (N = 19) | 0.20075 (0.20456) [lower limit 0.20456]
  24 Hours (N = 18) | 0.16325 (0.08983) [lower limit 0.08983]
  168 Hours (N = 2) | 0.05767 (NA) — Not calculated, insufficient samples

2. Primary Outcome: Summary of Pharmacokinetic Parameters Following Ivermectin Application.
Description: Plasma concentrations of ivermectin were measured by validated and appropriate bioanalytical instruments and methods before application and on Day 1 (0.5, 1, and 6 hours post-application), Day 2 (24 hours post-application), Day 8 (7 days post-application), and Day 15 (14 days post-application).
Time Frame: Before; 0.5, 1, 6, 24 hours, Day 8 and Day 15 post-application
Population: Plasma concentrations of Ivermectin were assessed in the pharmacokinetic (PK) population.
Measure: Mean (Standard Deviation); unit: ng/h/mL
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 20
ng/h/mL
  Time Averaged Plasma Concentration | 0.08708 (0.11102) [lower limit 0.11102]
  Area Under Plasma Concentration Last | 6.701 (11.23) [lower limit 11.23]
  Area Under Plasma Concentration 0 to 24 | 3.972 (3.5142) [lower limit 3.5142]

3. Secondary Outcome: Number of Participants Reporting Adverse Events Following Ivermectin Treatment
Description: Adverse events were assessed at each visit and during the follow up phone call on Day 28.
Time Frame: Day 1 up Day 28 post-application
Population: Adverse events were assessed in the intent-to-treat population.
Measure: Number; unit: Participants
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 30
Participants
  Diarrhea | 1
  Severe Diarrhea | 0
  Vomiting | 1
  Severe Vomiting | 0
  Gastroenteritis | 1
  Severe Gastroenteritis | 0
  Nasopharyngitis | 2
  Severe Nasopharyngitis | 0
  Upper Respiratory Tract Infection | 2
  Severe Upper Respiratory Tract Infection | 0
  Alanine Aminotransferase Increased | 2
  Severe Alanine Aminotransferase Increased | 0
  Aspartate Aminotransferase Increased | 1
  Severe Aspartate Aminotransferase Increased | 0
  Dehydration | 1
  Severe Dehydration | 0
  Dermatitis Diaper | 1
  Severe Dermatitis Diaper | 0
  Erythema | 5
  Severe Erythema | 0
  Pruritus | 1
  Severe Pruritus | 0

4. Secondary Outcome: Percentage of Participants Who Were Lice-Free by Visit Post-treatment With Ivermectin.
Description: Eradication of live lice was assessed by visual examination of the scalp and hair.
Time Frame: Day 2, Day 8 and Day 15 post-application
Population: Eradication of live lice was assessed in the intent-to-treat population.
Measure: Number; unit: Percent of Participants
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 30
Percent of Participants
  Day 2 (N = 30) | 97
  Day 8 (N = 29) | 90
  Day 15 (N = 28) | 89

5. Secondary Outcome: Percentage of Participants Who Were Lice-Free by Day 2 That Were Maintained Through Day 8 and Day 15 Post-treatment With Ivermectin.
Description: Eradication of live lice was assessed by visual examination of the scalp and hair before and following application of Ivermectin.
Time Frame: Day 2, Day 8 and Day 15 post-application
Population: Eradication of live lice was assessed in the intent to treat population.
Measure: Number; unit: Percent of Participants
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 30
Percent of Participants
  Eradication by Day 2 (N = 30) | 97
  Eradication Maintained Through Day 8 and 15 (N=29) | 86

6. Secondary Outcome: Liver Function Test Results at Before (Day 1) and Following Ivermectin Application on Days 2, 8, and 15 Post-application
Description: Liver function tests (Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, and Lactate Dehydrogenase) were performed before Ivermectin application on Day 1 (baseline) and on Days 2, 8, and 15 after application.
Time Frame: Day 1, Day 2, Day 8 and Day 15 post-application
Population: Liver function tests were performed in the intent to treat population.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 30
U/L
  Alkaline Phosphatase - Day 1 | 257.9 (59.5)
  Alkaline Phosphatase Day 2 | 258.0 (58.4)
  Alkaline Phosphatase Change from Day 1 to 2 | 4.2 (16.5)
  Alkaline Phosphatase Day 8 | 259.1 (51.0)
  Alkaline Phosphatase Change from Day 1 to 8 | -2.2 (28.4)
  Alkaline Phosphatase Day 15 | 258.3 (52.6)
  Alkaline Phosphatase Change from Day 1 to 15 | -2.9 (32.3)
  Alanine Aminotransferase Day 1 | 25.0 (20.5)
  Alanine Aminotransferase Day 2 | 25.7 (20.9)
  Alanine Aminotransferase Change from Day 1 to 2 | 0.2 (20.9)
  Alanine Aminotransferase Day 8 | 25.1 (22.1)
  Alanine Aminotransferase Change from Day 1 to 8 | -0.2 (5.3)
  Alanine Aminotransferase Day 15 | 24.1 (15.5)
  Alanine Aminotransferase Change from Day 1 to 15 | -1.1 (8.9)
  Aspartate Aminotransferase Day 1 | 42.6 (15.4)
  Aspartate Aminotransferase Day 2 | 41.1 (11.5)
  Aspartate Aminotransferase Change from Day 1 to 2 | -2.0 (15.4)
  Aspartate Aminotransferase Day 8 | 40.3 (14.0)
  Aspartate Aminotransferase Change from Day 1 to 8 | -2.3 (6.8)
  Aspartate Aminotransferase Day 15 | 39.5 (9.6)
  Aspartate Aminotransferase Change from Day 1 to 15 | -2.7 (10.2)
  Lactate Dehydrogenase Day 1 | 308.0 (87.5)
  Lactate Dehydrogenase Change Day 2 | 295.2 (35.8)
  Lactate Dehydrogenase Change from Day 1 to 2 | -16.8 (95.1)
  Lactate Dehydrogenase Day 8 | 295.1 (54.0)
  Lactate Dehydrogenase Change from Day 1 to 8 | -10.7 (80.2)
  Lactate Dehydrogenase 15 | 294.5 (61.3)
  Lactate Dehydrogenase Change from Day 1 to 15 | -9.2 (69.0)

7. Secondary Outcome: Liver Function Test Results at Before (Baseline) and Following Ivermectin Application on Days 2, 8, and 15 Post-application
Description: Liver function test (total bilirubin) was performed before treatment Day 1 (baseline) and following Ivermectin application on Days 2, 8, and 15 Post-application, respectively.
Time Frame: Day 1, Day 2, Day 8 and Day 15 post-application
Population: Liver function tests were performed in the intent to treat population.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 30
mg/dL
  Total Bilirubin - Day 1 | 0.3 (0.3)
  Total Bilirubin Day 2 | 0.3 (0.3)
  Total Bilirubin Change from Day 1 to 2 | -0.0 (0.1)
  Total Bilirubin Day 8 | 0.3 (0.3)
  Total Bilirubin Change from Day 1 to 8 | -0.0 (0.1)
  Total Bilirubin Day 15 | 0.3 (0.3)
  Total Bilirubin Change from Day 1 to 15 | -0.1 (0.2)

8. Primary Outcome: Summary of Pharmacokinetic Parameter (Mean Concentration) Following Ivermectin Application.
Description: as for outcome 2
Time Frame: Before; 0.5, 1, 6, 24 hours, Day 8 and Day 15 post-application
Population: Plasma concentrations of Ivermectin were assessed in the pharmacokinetic (PK) population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 20
ng/mL | 0.241 (0.23372)

9. Primary Outcome: Summary of Pharmacokinetic Parameter (Time of Observed Maximum Plasma Concentration) Following Ivermectin Application.
Description: as for outcome 2
Time Frame: Before; 0.5, 1, 6, 24 hours, Day 8 and Day 15 post-application
Population: Plasma concentrations of Ivermectin were assessed in the pharmacokinetic (PK) population.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 0.5% Ivermectin
Number analyzed (Participants) | 20
hour | 15.9 (10)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the day of application (Day 1) through Day 28 post-application
Arm/Group | 0.5% Ivermectin
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 11/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5% Ivermectin (N=30)
Gastroenteritis (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.5% Ivermectin (N=30)
Nasopharyngitis (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Alanine Aminotransferase Increased (Investigations) | 2
Erythema (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications